CLINICAL TRIAL: NCT00951379
Title: Phase IIB Randomized, Placebo Controlled Trial of Pioglitazone for Oral Premalignant Lesions an Inter-consortium Collaborative Study
Brief Title: Pioglitazone for Oral Premalignant Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-03152; NCI-2012-03152 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UWI H-2009-0106; MDA-2009-0339 (Other: MD Anderson Cancer Center (MDACC)); INC07-10-01 (Other: DCP); N01CN35159 (NIH); N01CN35153 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2014-06

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Pioglitazone Hydrochloride) (Experimental): Three (3) Pioglitazone 15 mg capsules by mouth once daily for 24 weeks
  Interventions: Drug: Pioglitazone hydrochloride; Other: laboratory biomarker analysis
- Arm II (Placebo) (Placebo Comparator): Three (3) placebo capsules by mouth once daily for 24 weeks
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Pioglitazone hydrochloride — Three (3) pioglitazone 15 mg capsules by mouth once daily for 24 weeks (+/- 1 week)
  Other Names: Actos; pioglitazone
  Arms: Arm I (Pioglitazone Hydrochloride)
Other: placebo — Three (3) pioglitazone placebo capsules by mouth once daily for 24 weeks (+/- 1 week)
  Other Names: PLCB
  Arms: Arm II (Placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The goal of this clinical research study is to learn how Actos (pioglitazone) may affect oral premalignant lesions (OPLs) and/or the risk of mouth cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical and histologic response of oral premalignant lesions to 24 weeks of therapy with pioglitazone, 45 mg once daily (qd), defined as 50% or greater reduction in the sum of all measured products of perpendicular dimensions of target lesions, or improvement in the degree of dysplasia or hyperplasia.

SECONDARY OBJECTIVES:

I. To determine the degree of change of putative biomarkers of pioglitazone efficacy including (but not restricted to) and in order of priority, tissue levels of:

* PPAR gamma,
* cyclin D1 and p21 as indirect measures of pharmacological effect
* TUNEL for apoptosis and Ki-67 for proliferation
* transglutaminase and involucrin as markers of squamous differentiation
* 15-PGDH, loss of heterozygosity (LOH). II. To determine the degree of change of C-reactive protein (CRP) in plasma. III. To assess tobacco and alcohol use among trial participants and to examine the relationship of tobacco and alcohol use to treatment response.

IV. To assess the safety of this agent in this population.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pioglitazone hydrochloride orally (PO) once daily (QD) for 24 weeks.

ARM II: Patients receive placebo PO QD for 24 weeks.

After completion of study treatment, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* STAGE I:
* Males or females with a suspected or histologically confirmed oral premalignant lesion(s) (up to three target lesions may be followed for the purpose of the study) that has a length (longest diameter) of 8 mm or greater and width (diameter perpendicular to greatest length) of 3 mm or greater in size

  * If a participant has had a biopsy of the target oral premalignant lesions (OPL) lesion(s) within 6 weeks prior to the screening visit and archival tissue is available and the participant agrees to have archival tissue used for histologic confirmation and biomarker analysis, then NO additional biopsies (of the OPL) need to be performed at the screening visit; the pre-screening biopsy must undergo centralized pathology review before the second stage of registration can be performed; if archival tissue is not available, a waiting period of 6 weeks from the time of the last biopsy must be observed before re-biopsy for study purposes
  * If a participant has not had a biopsy of the suspected OPL at the time of the screening visit, then a biopsy of the lesion must be performed during the screening visit; the screening biopsy must undergo centralized pathology review before the second stage of registration can be performed
* The participant's life expectancy is > 6 months
* The participant has discontinued any other oral cancer chemopreventive therapy at least 12 weeks prior to the baseline visit and all toxicities have been fully resolved; daily aspirin is permitted
* The participant is willing and able to fully participate for the duration of the study
* Women must not be pregnant or lactating; women of child-bearing potential (women are considered not of childbearing potential if they are at least two years postmenopausal and/or surgically sterile) must have used adequate contraception (abstinence; barrier methods such as IUD, diaphragm with spermicidal gel, condom, or others; and hormonal methods such as birth control pills or others) since her last menses prior to study entry; women of child-bearing potential and men must agree to use adequate contraception for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* STAGE II:
* The participant has one or more target lesions histologically confirmed by a biopsy obtained no more than 9 weeks prior to randomization, that is either:

  * An EARLY premalignant lesion defined to be at high risk:

    * Mild dysplasia of any site
    * Hyperplastic leukoplakia of a high-risk site

      * Dorsal, lateral or ventral tongue
      * Floor of mouth
  * An ADVANCED premalignant lesion defined as the presence of at least one of the following:

    * Moderate dysplasia
    * Severe dysplasia (excluding carcinoma in situ)
    * Erythroplakia (due to the high risk for progression associated with erythroplakia, erythroplakia of any histology will be defined as an ADVANCED oral premalignant lesion)
* Hemoglobin levels equal to or above the lower limit of normal
* White blood cells >= 3,000/uL
* Platelets >= 125,000/uL
* Total bilirubin =< 1.5 * upper limit of normal (ULN)
* BUN and serum creatinine =< 1.5 * ULN
* Glucose, serum < 200 mg/dL
* The participant's Eastern Cooperative Oncology Group (ECOG) performance status is 0 or 1
* If the participant is female and of childbearing potential and not lactating she has a documented negative serum pregnancy test within 14 days prior to randomization
* The participant has a baseline EKG that does not show signs of acute cardiac ischemia or cardiac dysrhythmia (except for 1st degree AV block or chronic atrial fibrillation); EKG can be an earlier report within 12 weeks prior to registration
* Participants using the drugs listed below may not be randomized unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 3 days prior to starting pioglitazone or placebo on this study; the use of the following drugs or drug classes is prohibited during pioglitazone/placebo treatment: participants taking inhibitors of CYP2C8 (gemfibrozil, ketoconazole, quercetin, trimethoprim), enzyme inducers of CYP2C8 (cortisol, dexamethasone, phenobarbital, rifampin), and CYP3A4 substrate

Exclusion Criteria:

* The participant has active cancer or carcinoma in situ of the head and neck
* The participant has a contraindication to biopsy
* The participant has presence of congestive heart failure (New York Heart Association (NYHA) class II-IV), uncontrolled hypertension (systolic > 150 or diastolic > 100), or unstable angina
* The participant has any history of congestive heart failure or history of myocardial infarction within the past 6 months
* The participant exhibits clinical evidence of active liver disease or history of chronic liver disease
* The participant has > Common Terminology Criteria for Adverse Events (CTCAE) grade 1 edema
* The participant has known diabetes and is on insulin or oral agents; the participant is receiving medical therapy for dysregulated blood sugar
* The participant who currently receives an enzyme inhibitor of CYP2C8 (gemfibrozil, ketoconazole, quercetin, trimethoprim), or enzyme inducer of CYP2C8 (cortisol, dexamethasone, phenobarbital, rifampin), or CYP3A4 substrate will not be eligible for randomization after assessing eligibility in stage two unless he/she will not be eligible for randomization after assessing eligibility in stage two unless he/she is willing to stop these drugs and possibly replace them with alternative therapies
* The participant currently receives pregabalin or thioridazine
* The participant has experienced jaundice with Rezulin (troglitazone)
* The participant has a history of colorectal cancer, familial adenomatous polyposis (FAP) or hereditary non-polyposis colorectal cancer (HNPCC)
* The participant has a history of bladder cancer or in situ bladder cancer
* The participant has a history of invasive cancer within the past 18 months (excluding non-melanoma skin cancer and in situ cervical cancer); participants (excluding those with a history of colorectal cancer, FAP, HNPCC, bladder cancer or in situ bladder cancer) who received curative treatment and have shown no evidence of recurrence for 18 months will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Powel H. Brown, Principal Investigator — University of Texas MD Anderson Cancer Center, Consortium PI
Locations (13):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- BC Cancer Agency (Vancouver Cancer Centre), Vancouver, British Columbia, Canada
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Gates JC, Abouyared M, Shnayder Y, Farwell DG, Day A, Alawi F, Moore M, Holcomb AJ, Birkeland A, Epstein J. Clinical Management Update of Oral Leukoplakia: A Review From the American Head and Neck Society Cancer Prevention Service. Head Neck. 2025 Feb;47(2):733-741. doi: 10.1002/hed.28013. Epub 2024 Nov 25. PMID 39584361
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org
- See also: National Cancer Institute (NCI) Central Website for Cancer Research — http://www.cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: first participant accrued July 12, 2010 and the last participant accrued on September 10, 2013. Recruitment done in medical clinic settings across the United States, at the European Institute of Oncology in Milan, Italy, and at the BC Cancer Center, Vancouver, British Columbia, Canada.
Pre-assignment Details: Of the 99 participants screened during recruitment phase, 47 participants failed screening and were excluded from the trial before assignment to groups. Due to slow accrual, the study was terminated in September 2013.
Period: Overall Study
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Started | 27 | 25
Completed | 21 | 23
Not Completed | 6 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (8.3) | 59.0 (10.3) | 59.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45
  Italy | 4 | 3 | 7
Alcohol Use at Baseline [Number; unit: participants] — Heavy drinkers are participants who drank every day; Light drinkers are participants who drank on some days; Non-drinkers are former drinkers or those who never drank alcohol.
  participants
    Heavy | 2 | 3 | 5
    Light | 17 | 17 | 34
    Non-Drinker | 8 | 5 | 13
Smoking Use at Baseline [Number; unit: participants]
  Current | 6 | 6 | 12
  Former | 12 | 7 | 19
  Never | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response <Clinical and Histologic Response Defined as 50% or Greater Reduction in the Sum of the Measured Products of Perpendicular Dimensions of the Target Lesion(s) or Improvement in the Degree of Dysplasia or Hyperplasia>
Description: Overall Dichotomized Clinical and Histologic Response defined as 50% or greater reduction in sum of the measured products of perpendicular dimensions of the target lesion(s) or improvement in the degree of dysplasia or hyperplasia where complete (CR) or partial response (PR) in either clinical or histologic outcome assessed according to criteria given recorded as Response or No Response and analyzed as a dichotomous variable. Clinical Response = CR: Disappearance all evidence target & non-target lesions; PR: >/=50% reduction in sum products of diameters all target lesion(s). Non-target lesions may not increase >/=25% in size & no new lesion. Histologic Response = CR: Complete reversal of dysplasia or hyperplasia to normal epithelium in all biopsied lesions. PR: Improvement of degree of dysplasia or hyperplasia in all biopsied lesion(s) from advanced to early, or from early to normal epithelium in some lesions while other biopsied lesions remain stable.
Time Frame: Response assessed at Week 24 ±1 Week
Population: All participants who received at least one dose of treatment. One participant in the Pioglitazone arm never received study drug.
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 25
participants
  Response | 12 | 8
  No Response | 14 | 17

2. Secondary Outcome: Number of Participants With >5.0 mg/L in Level of C-reactive Protein in Plasma
Description: Degree of change of C-reactive protein (CRP) in plasma serum via blood tests.
  The longitudinal regression models for analysis of the change in CRP in plasma used, with suitable transformation if necessary to satisfy the model assumptions, with treatment, stage and biomarker value at screening visit as covariates.
Time Frame: Baseline to end of study, 24 weeks
Population: Pioglitazone's 26 had 24 evaluable specimens at baseline & 20 evaluable at end of study with 2 of those not available for CRP>5 baseline measure: Placebo's 25 had 25 evaluable specimens at baseline & 21 at end of study. Analysis based on specimen viability/availability, no exclusions made for other reasons, participant needed 1/+ dose of treatment.
Measure: Number; unit: participants
Groups:
- Pioglitazone: CRP>5 at Baseline: Measure at baseline, followed by Pioglitazone treatment three 15 mg capsules orally/day for 24 weeks
- Pioglitazone: CRP>5 End of Study: Measure at end of Pioglitazone treatment, approximately 24 weeks
- Placebo: CRP> 5 Baseline: Measure at baseline, followed by Placebo treatment three capsules orally/day for 24 weeks
- Placebo: CRP>5 End of Study: Measure at end of Placebo treatment, approximately 24 weeks
Arm/Group | Pioglitazone: CRP>5 at Baseline | Pioglitazone: CRP>5 End of Study | Placebo: CRP> 5 Baseline | Placebo: CRP>5 End of Study
Number analyzed (Participants) | 24 | 20 | 25 | 21
participants
  Yes | 6 | 1 | 4 | 4
  No | 18 | 19 | 21 | 17

3. Secondary Outcome: Number of Participants With Level of C-reactive Protein in Plasma Decrease From >5.0 mg/L to <= 5.0 mg/L From Baseline to End of Study
Description: The longitudinal regression models for analysis of the change in CRP in plasma will be used, with suitable transformation if necessary to satisfy the model assumptions, with treatment, stage and biomarker value at screening visit as covariates.
Time Frame: Baseline to end of study, 24 weeks
Population: Pioglitazone's 26 had 20 evaluable specimens at baseline & 20 at end of study with 2 of those not available for the CRP>5 baseline measure & Placebo's 25 had 25 evaluable at baseline & 21 evaluable at end of study. Analysis based on specimen viability/availability, no exclusions made for other reasons, participants needed 1/+ dose of treatment.
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 18 | 21
participants
  Yes | 3 | 0
  No | 15 | 21

4. Secondary Outcome: Number of Participant With Clinical Response by Baseline Characteristics: Tobacco Use
Description: Tobacco use summarized by treatment stratified by stage and by group. In addition, the effects of tobacco and alcohol use on the primary endpoint of clinical response assessed.
Time Frame: Up to 26 weeks
Population: Analysis includes all participants who received at least one dose of treatment. One participant in the Pioglitazone arm never received study drug.
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 25
participants
  Never Smoked | 4 | 5
  Former Smoker | 5 | 2
  Current Smoker | 2 | 1

5. Secondary Outcome: Number of Participant With Clinical Response by Baseline Characteristics: Alcohol Use
Description: Alcohol use will be summarized by treatment stratified by stage and by group. In addition, the effects of tobacco and alcohol use on the primary endpoint of clinical and pathological response assessed using statistical regression models in an exploratory fashion. Heavy drinkers are participants who drank every day; Light drinkers are participants who drank on some days; Non-drinkers are former drinkers or those who never drank alcohol.
Time Frame: Up to 26 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 25
participants
  Non-Drinker | 2 | 2
  Light Drinker | 8 | 6
  Heavy Drinker | 1 | 0

6. Secondary Outcome: Number of Participants Affected by Adverse Events Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4.0)
Description: All adverse events (including serious) and clinical laboratory toxicity summarized affected organ system. Reporting based on the NCI CTCAE v4.0 by treatment, details included in later Adverse Event Module of results.
Time Frame: Up to 26 weeks
Population: Population includes all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 27 | 25
participants
  Blood & Lymphatic System Disorders | 1 | 0
  Cardiac Disorders | 3 | 2
  Ear & Labyrinth Disorders | 0 | 2
  Eye Disorders | 7 | 2
  Gastrointestinal Disorders | 23 | 22
  General Disorders & Administration Site Conditions | 12 | 10
  Infections and Infestations | 9 | 8
  Injury, Poisoning and Procedural Complications | 0 | 2
  Investigations | 3 | 2
  Metabolism and Nutrition Disorders | 2 | 0
  Musculoskeletal and Connective Tissue Disorders | 7 | 8
  Neoplasms Benign, Malignant and Unspecified | 1 | 0
  Nervous System Disorders | 14 | 7
  Psychiatric Disorders | 3 | 1
  Reproductive System and Breast Disorders | 1 | 0
  Respiratory, Thoracic and Mediastinal Disorders | 18 | 9
  Skin and Subcutaneous Tissue Disorders | 4 | 2
  Surgical and Medical Procedures | 2 | 3
  Vascular Disorders | 5 | 12

7. Secondary Outcome: Biomarker Measurements at Scheduled Visits: Tissue Levels of Cyclin D1
Description: Tissue levels of Cyclin D1 as indirect measures of pharmacological effect assessed by immunohistochemistry (IHC). Tissue levels of biomarkers assessed from the biopsy obtained at the Screening Clinic Visit and Week 24 ± 1 Week, and plasma levels of biomarkers assessed from blood collected at the Baseline Clinic Visit and Week 24 ± 1 Week. Data reported as percentage of cells staining positive, according to nuclear or cytoplasmic compartments.
Time Frame: Baseline to end of study, 24 weeks
Population: Two participants in the Pioglitazone arm were not analyzed for Cyclin D1 end of study score. Analysis is based on specimen viability/availability. No exclusions are made for any other reason.
Measure: Mean (Standard Deviation); unit: percentage of staining cells positive
Groups:
- Pioglitazone: Baseline: Measure at baseline, followed by Pioglitazone treatment three 15 mg capsules orally/day for 24 weeks
- Pioglitazone: End of Study: Measure at end of Pioglitazone treatment, approximately 24 weeks
- Placebo: Baseline: Measure at baseline, followed by Placebo treatment three capsules orally/day for 24 weeks
- Placebo: End of Study: Measure at end of Placebo treatment, approximately 24 weeks
Arm/Group | Pioglitazone: Baseline | Pioglitazone: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 25 | 23 | 24 | 24
percentage of staining cells positive | 15.5 (10.0) | 12.7 (6.9) | 12.8 (7.9) | 12.9 (7.0)

8. Secondary Outcome: Biomarker Measurements at Scheduled Visits: Tissue Levels of Ki-67
Description: Tissue levels of Ki-67 for proliferation assessed by immunohistochemistry (IHC). Tissue levels of biomarkers assessed from the biopsy obtained at the Screening Clinic Visit and Week 24 ± 1 Week, and plasma levels of biomarkers assessed from blood collected at the Baseline Clinic Visit and Week 24 ± 1 Week. Data reported as percentage of cells staining positive, according to nuclear or cytoplasmic compartments.
Time Frame: Baseline to end of study, 24 weeks
Population: Four participants in the Pioglitazone arm were not analyzed for Ki-67 end of study score. Analysis is based on specimen viability/availability. No exclusions are made for any other reason.
Measure: Mean (Standard Deviation); unit: percentage of staining cells positive
Arm/Group | Pioglitazone: Baseline | Pioglitazone: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 25 | 21 | 24 | 24
percentage of staining cells positive | 9.2 (4.6) | 8.9 (4.2) | 10.7 (6.5) | 8.2 (4.6)

9. Secondary Outcome: Biomarker Measurements at Scheduled Visits: Tissue Levels of p21
Description: Tissue levels of p21 as indirect measures of pharmacological effect assessed by immunohistochemistry (IHC). Tissue levels of biomarkers assessed from the biopsy obtained at the Screening Clinic Visit and Week 24 ± 1 Week, and plasma levels of biomarkers assessed from blood collected at the Baseline Clinic Visit and Week 24 ± 1 Week. Data reported as percentage of cells staining positive, according to nuclear or cytoplasmic compartments.
Time Frame: Baseline to end of study, 24 weeks
Population: Two participants in the Pioglitazone arm were not analyzed for p21 end of study score. Analysis is based on specimen viability/availability. No exclusions are made for any other reason.
Measure: Mean (Standard Deviation); unit: percentage of staining cells positive
Arm/Group | Pioglitazone: Baseline | Pioglitazone: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 25 | 23 | 24 | 24
percentage of staining cells positive | 18.7 (10.2) | 19.3 (10.6) | 17.7 (10.8) | 15.6 (7.4)

10. Secondary Outcome: Biomarker Measurements at Scheduled Visits: Tissue Levels of B-cell Lymphoma 2 (Bcl2)
Description: Tissue levels of Bcl2 as indirect measures of pharmacological effect assessed by immunohistochemistry (IHC). Tissue levels of biomarkers assessed from the biopsy obtained at the Screening Clinic Visit and Week 24 ± 1 Week, and plasma levels of biomarkers assessed from blood collected at the Baseline Clinic Visit and Week 24 ± 1 Week. Data reported a percentage of cells staining positive, according to nuclear or cytoplasmic compartments.
Time Frame: Baseline to end of study, 24 weeks
Population: Four participants of 25 overall in the Pioglitazone arm were not analyzed for Bcl2 end of study score and one participant in Placebo was not analyzed for Bcl2 baseline score. Analysis is based on specimen viability/availability. No exclusions are made for any other reason.
Measure: Mean (Standard Deviation); unit: percentage of staining cells positive
Arm/Group | Pioglitazone: Baseline | Pioglitazone: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 25 | 21 | 23 | 24
percentage of staining cells positive | 2.8 (3.2) | 2.3 (2.3) | 4.2 (5.0) | 4.6 (8.3)

11. Secondary Outcome: Biomarker Measurements at Scheduled Visits: Tissue Levels of PPARG Nucleus and PPARG Cytoplasm
Description: Tissue levels of Peroxisome proliferator-activated receptor gamma (PPARG) Nucleus and PPARG Cytoplasm as indirect measures of pharmacological effect, PPAR gamma assessed by immunohistochemistry. Tissue levels of biomarkers assessed from the biopsy obtained at the Screening Clinic Visit and Week 24 ± 1 Week, and plasma levels of biomarkers assessed from blood collected at the Baseline Clinic Visit and Week 24 ± 1 Week. Data reported as percentage of cells staining positive, according to nuclear or cytoplasmic compartments.
Time Frame: Baseline to end of study, 24 weeks
Population: Four participants in the Pioglitazone arm were not analyzed at end of study, and two participants in Placebo were not analyzed for PPARG baseline scores. Analysis is based on specimen viability/availability. No exclusions are made for any other reason.
Measure: Mean (Standard Deviation); unit: percentage of staining cells positive
Arm/Group | Pioglitazone: Baseline | Pioglitazone: End of Study | Placebo: Baseline | Placebo: End of Study
Number analyzed (Participants) | 25 | 21 | 22 | 24
percentage of staining cells positive
  PPARG Nucleus | 10.8 (15.7) | 7.3 (7.5) | 12.4 (10.4) | 6.8 (7.2)
  PPARG Cytoplasm | 21.7 (25.8) | 23.5 (28.0) | 20.2 (29.9) | 21.5 (31.3)

12. Primary Outcome: Dichotomized Histologic Response (HR): Participant Complete or Partial Response Defined as =/>50% Reduction in the Sum of the Measured Products of Perpendicular Dimensions of the Target Lesion(s) or Improvement in the Degree of Dysplasia or Hyperplasia
Description: HR according to criteria & recorded as Response or No Response, analyzed as dichotomous variable. CR: Complete reversal dysplasia/hyperplasia to normal epithelium in all biopsied lesions. PR: Improvement of degree dysplasia/hyperplasia in all biopsied lesion from advanced to early, or from early to normal epithelium in some lesions while other biopsied lesions remain stable. No Change (NC): No change in degree dysplasia/hyperplasia in all biopsied lesions, anything not CR, PR or PD. Progressive Disease (PD): Any increase in severity histology grade any biopsied lesion. Early premalignant lesion: lesion defined high risk, indicated by presence of one: hyperplasia at high-risk sites (dorsal, lateral or ventral tongue, or floor of mouth) ONLY, or mild dysplasia. Advanced premalignant lesion: lesion with presence of one: moderate dysplasia or severe dysplasia (excluding CIS), erythroplakia with hyperplasia or of any severity of dysplasia.
Time Frame: Response assessed at Week 24 ±1 Week
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 25
participants
  Response | 2 | 2
  No Response | 24 | 23

13. Primary Outcome: Dichotomized Clinical Response: Participant Complete or Partial Response Defined as =/>50% Reduction in the Sum of the Measured Products of Perpendicular Dimensions of the Target Lesion(s) or Improvement in the Degree of Dysplasia or Hyperplasia
Description: Clinical Response assessed according to criteria & recorded as Response or No Response, analyzed as dichotomous variable. Complete Response (CR): Disappearance of all evidence of target AND non-target lesions. Partial Response (PR): greater than or equal to 50% reduction in the sum of the products of diameters of all target lesion(s). Non-target lesions may not increase greater than or equal 25% in size and no new lesion may appear. No Change (NC): No change in the size of the lesion(s) and no new lesions appearing, i.e. anything that is not CR, PR or PD. Progressive Disease (PD): Any increase greater than or equal to 25% in the product of the diameters of any measurable lesions or in the estimated size of non-measurable lesions or the appearance of an unequivocal new lesion.
Time Frame: Response assessed at Week 24 ±1 Week
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 26 | 25
participants
  Response | 11 | 8
  No Response | 15 | 17

ADVERSE EVENTS:
Time Frame: Adverse signs and symptoms recorded at each clinic visit beginning week 4 through week 24 (± 1 week). All adverse events followed according to established standards of care. Overall study period: May 2010 to March 2014.
Description: Study source vocabulary for the study began as CTCAE version 3.0 and was translated to version 4.0.
Arm/Group | Arm I (Pioglitazone Hydrochloride) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 3/27 | 1/25
Other Adverse Events (participants affected / at risk) | 22/27 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pioglitazone Hydrochloride) (N=27) | Arm II (Placebo) (N=25)
heart failure (Cardiac disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
laparoscopic hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — Total laparoscopic hysterectomy with bilateral salpingo-oophorectomy, sacrocolpopexy and midurethral tissue fixation system sling
Pre-existing abdominal aortic aneurysm (Surgical and medical procedures) | 0 (0) | 1 (1) — hospitalization for repair of pre-existing abdominal aortic aneurysm
right femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pioglitazone Hydrochloride) (N=27) | Arm II (Placebo) (N=25)
anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
palpitations (Cardiac disorders) | 2 (2) | 0 (0)
hearing issues (Ear and labyrinth disorders) | 0 (0) | 1 (1)
hearing loss, earwax (Ear and labyrinth disorders) | 0 (0) | 1 (1)
bilateral burning eye (Eye disorders) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 1 (1) | 1 (1)
conjunctival abrasion (Eye disorders) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
myopia (Eye disorders) | 1 (1) | 0 (0)
red bloodshot eyes (Eye disorders) | 1 (1) | 0 (0)
scotoma of right eye (Eye disorders) | 1 (1) | 0 (0)
vitreous detachment of left eye (Eye disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
lump under tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
oral pain (Gastrointestinal disorders) | 6 (11) | 4 (4)
periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
striations on tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
red spots right lower lip (Gastrointestinal disorders) | 1 (1) | 0 (0)
stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
edema limbs (General disorders) | 2 (2) | 2 (2)
facial pain (General disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 3 (3) | 4 (5)
flu like symptoms (General disorders) | 2 (2) | 1 (1)
malaise (General disorders) | 2 (2) | 1 (1)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
sluggishness (General disorders) | 1 (1) | 0 (0)
suddenly famished (General disorders) | 1 (1) | 0 (0)
bladder infection (Infections and infestations) | 0 (0) | 1 (1)
bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
toe infection (Infections and infestations) | 0 (0) | 1 (1)
lip infection (Infections and infestations) | 0 (0) | 1 (1)
lung infection (Infections and infestations) | 1 (1) | 1 (1)
sinusitis (Infections and infestations) | 1 (1) | 1 (1)
skin infection (Infections and infestations) | 1 (1) | 0 (0)
soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
thrush in throat (Infections and infestations) | 1 (1) | 0 (0)
tooth infection (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
alanine aminotransferase (ALT) Increased (Investigations) | 0 (0) | 1 (1)
creatinine increased (Investigations) | 1 (1) | 0 (0)
weight gain (Investigations) | 1 (1) | 0 (0)
weight loss (Investigations) | 1 (1) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
increased chloride (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arms burning sensaton (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
mild leg cramps at night (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle pain right hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
rotator cuff trauma resulting from a fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 3 (3) | 2 (2)
dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 5 (7) | 2 (2)
hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
sinus pain (Nervous system disorders) | 1 (1) | 1 (1)
somnolence (Nervous system disorders) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 1 (1) | 1 (2)
anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
dry nasal passages (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
slight metallic smell (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
bee sting (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
skin dyschromia of arms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
small non-painful reddened area lower left arm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
keratotic horns on head (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
molar extracted due to failed root canal (Surgical and medical procedures) | 0 (0) | 1 (1)
outpatient surgery, knee meniscus repair (Surgical and medical procedures) | 0 (0) | 1 (1)
trans oral surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 4 (6) | 11 (14)
minor venous insufficiency of the legs (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less